CLINICAL TRIAL: NCT06107504
Title: Prevention of Post-sphincterotomy Bleeding by Endoscopic Tranexamic Acid and Sucralfate Administration: A Randomized Controlled Trial
Brief Title: Prevention of Post-sphincterotomy Bleeding
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Hsueh-Chien Chiang, Principal Investigator, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B-BR-112-038
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2024-12

CONDITIONS: Post-ERCP Bleeding
MeSH Terms: interventions — Sucralfate; Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Participants will be recruited from the volunteers with choledocholithiasis at National Cheng Kung University Hospital and Siriraj Hospital. Eligible participants include patients aged ≥ 18 years who accept ERCP and sphincterotomy for common bile duct (CBD) stone extraction. Patient consent forms will be given and explained to all patients before the ERCP. Exclusion criteria include patients with no schedules for sphincterotomy, unsuccessful CBD cannulation, and allergy to sucralfate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): After the EST and stone extraction, we will randomly assign the patients to either a control or an intervention group. After EST, if immediate bleeding occurs, we will apply standard endoscopic therapy by either local injection of diluted epinephrine or heater probe coagulation. After then, we will spray 1g of sucralfate powder and 0.5g of tranexamic acid powder through a duodenoscope precisely on the EST wound in the intervention group.
  Interventions: Drug: Sucralfate
- Control group (No Intervention): After the EST and stone extraction, we will randomly assign the patients to either a control or an intervention group. After EST, if immediate bleeding occurs, we will apply standard endoscopic therapy by either local injection of diluted epinephrine or heater probe coagulation.

INTERVENTIONS:
Drug: Sucralfate — 2g of sucralfate powder and 1g of tranexamic acid powder will be sprayed after EST
  Other Names: Tranexamic acid
  Arms: Intervention group

SUMMARY:
Background and Aim: Endoscopic retrograde cholangiopancreatography (ERCP) and sphincterotomy (EST) are standard treatments for choledocholithiasis. However, 10% of post-EST bleeding was reported. Currently, there are no effective methods or medications for the prevention of post-EST bleeding. This study aimed to investigate whether the local administration of TXA and sucralfate can reduce the post-EST bleeding event.

Methods: This is a randomized clinical trial. Patients with choledocholithiasis scheduled for ERCP with EST at National Cheng Kung University Hospital and Siriraj Hospital were enrolled. The study will recruit 120 patients. After randomization, 60 patients will be classified into the intervention group and 60 into the control group. The participants will receive standard ERCP and EST for common bile duct stone removal. If immediate polypectomy bleeding occurs, the investigators will apply standard endoscopic therapy by either local injection of diluted epinephrine or heater probe coagulation. After then, the investigators will spray 2g of sucralfate powder and 1g of tranexamic acid through duodenoscopy precisely on the post-EST wound in the intervention group. All enrolled patients will be monitored for delayed bleeding for 14 days after the ERCP.

DETAILED DESCRIPTION:
Endoscopic retrograde cholangiopancreatography (ERCP) is an advanced endoscopic procedure combining endoscopy and fluoroscopy to diagnose and treat diseases of the pancreaticobiliary ductal system, including choledocholithiasis, biliary strictures, and cholangitis. ERCP is associated with a higher rate of complications than other endoscopic procedures, including post-ERCP pancreatitis (PEP), bleeding, perforation, and biliary tract infection. The incidence rate of ERCP-related complications has been reported at approximately 10 percent, with mortality rates ranging from 0.1 to 1.4 percent. Despite recent technological advancements and safety precautions, the ERCP procedure-related death rates have remained high.

Among all complications, delayed bleeding after sphincterotomy (EST) is a nightmare for both clinical physicians and endoscopists. Post-EST bleeding results in Tarry-bloody stool and anemia, increasing the mortality rate and hospital stay. While non-steroidal anti-inflammatory drugs (NSAIDs), pancreatic stents, and intravenous fluids can help prevent post-ERCP pancreatitis, there is no effective methodology or medication for bleeding prevention currently. Therefore, developing a prevention method for post-EST bleeding is urgent and important.

Tranexamic acid (TXA) is a well-known antifibrinolytic agent that inhibits fibrin degradation by binding to tissue plasminogen, thereby preventing blood clot lysis and reducing bleeding. A recent study evaluating the effect of topical tranexamic acid (TXA) powder on bleeding peptic ulcers demonstrated that the precise endoscopic administration of TXA powder can enhance the stop-bleeding effect.

Sucralfate, a complex of aluminum hydroxide and sucrose octa sulfate, can bind to the wound base. This protective barrier can prevent the wound from further environmental injury. Sucralfate has been widely used for wounds and ulcer treatment, e.g., skin wounds, oral ulcers, and peptic ulcers. With the protective effect of the papilla mucosa, sucralfate can cover the EST wound and has the potential to avoid further environmental damage. In combination with TXA powder in stabilizing the clotting, we expect the post-EST bleeding event will reduce. Therefore, this study aimed to investigate whether the combination therapy of topical administration of TXA and sucralfate after EST can reduce the post-EST bleeding event.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years who accept ERCP and sphincterotomy for common bile duct (CBD) stone extraction

Exclusion Criteria:

* Paitnets with no schedules for sphincterotomy
* Paitnets with unsuccessful CBD cannulation
* Patients with allergy to sucralfate

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
The incident rate of delayed post-ERCP bleeding during the study period | 14 days
  The occurrence of delayed post-ERCP bleeding during the study period. Delayed post-ERCP bleeding was defined as remarkable hematochezia or Tarry stool with endoscopic evidence of post-EST wound bleeding.

SECONDARY OUTCOMES:
The incident rate of post-EST wound bleeding requiring transarterial embolization or emergency surgery | 14 days
  The incident rate of post-EST wound bleeding requiring transarterial embolization or emergency surgery.
The incidence rate of Hb loss > 2g/dL | 3 days
  The incidence rate of Hb loss > 2g/dL the day after ERCP
The mortality rate | 14 days
  All-cause mortality after EST
The incident rate post-ERCP pancreatitis | 14 days
  The incident rate post-ERCP pancreatitis after ERCP. The definition is epigastric pain and elevated lipase.
The Hb loss | 3 days
  The Hb decreased level during post-EST bleeding or day 2 after EST

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Other (Non U.s.), Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
IPD can be shared after publication

REFERENCES:
- [Background] ASGE Standards of Practice Committee; Buxbaum JL, Abbas Fehmi SM, Sultan S, Fishman DS, Qumseya BJ, Cortessis VK, Schilperoort H, Kysh L, Matsuoka L, Yachimski P, Agrawal D, Gurudu SR, Jamil LH, Jue TL, Khashab MA, Law JK, Lee JK, Naveed M, Sawhney MS, Thosani N, Yang J, Wani SB. ASGE guideline on the role of endoscopy in the evaluation and management of choledocholithiasis. Gastrointest Endosc. 2019 Jun;89(6):1075-1105.e15. doi: 10.1016/j.gie.2018.10.001. Epub 2019 Apr 9. PMID 30979521
- [Background] Fujita K, Yazumi S, Matsumoto H, Asada M, Nebiki H, Matsumoto K, Maruo T, Takenaka M, Tomoda T, Onoyama T, Kurita A, Ueki T, Katayama T, Kawamura T, Kawamoto H; Bilio-pancreatic Study Group of West Japan. Multicenter prospective cohort study of adverse events associated with biliary endoscopic retrograde cholangiopancreatography: Incidence of adverse events and preventive measures for post-endoscopic retrograde cholangiopancreatography pancreatitis. Dig Endosc. 2022 Sep;34(6):1198-1204. doi: 10.1111/den.14225. Epub 2022 Feb 4. PMID 34963021
- [Background] Akshintala VS, Sperna Weiland CJ, Bhullar FA, Kamal A, Kanthasamy K, Kuo A, Tomasetti C, Gurakar M, Drenth JPH, Yadav D, Elmunzer BJ, Reddy DN, Goenka MK, Kochhar R, Kalloo AN, Khashab MA, van Geenen EJM, Singh VK. Non-steroidal anti-inflammatory drugs, intravenous fluids, pancreatic stents, or their combinations for the prevention of post-endoscopic retrograde cholangiopancreatography pancreatitis: a systematic review and network meta-analysis. Lancet Gastroenterol Hepatol. 2021 Sep;6(9):733-742. doi: 10.1016/S2468-1253(21)00170-9. Epub 2021 Jun 30. PMID 34214449
- [Background] Leung WK, But DY, Wong SY, Tong TS, Liu KS, Cheung KS, Tsang SH, Chok KS, Poon RT, Hung IF. Prevention of post-sphincterotomy bleeding by proton pump inhibitor: A randomized controlled trial. J Dig Dis. 2018 Jun;19(6):369-376. doi: 10.1111/1751-2980.12604. Epub 2018 May 24. PMID 29722146
- [Background] Yu Z, He J, Cao R, Yang Z, Li B, Hong J, Chen Y, Zhu L. Proton pump inhibitor has no effect in the prevention of post-endoscopic sphincterotomy delayed bleeding: a prospective randomized controlled trial. Front Med (Lausanne). 2023 Jun 2;10:1179512. doi: 10.3389/fmed.2023.1179512. eCollection 2023. PMID 37332745
- [Background] Chiang HC, Chen PJ, Yang EH, Hsieh MT, Shih IC, Cheng HC, Chang WL, Chen WY, Chiu HC, Kuo HY, Tsai WC, Lo YN, Yang KC, Chiang CM, Chen WC, Huang KK, Tseng HH, Chen CY, Lin XZ, Chuang CH. Precise application of topical tranexamic acid to enhance endoscopic hemostasis for peptic ulcer bleeding: a randomized controlled study (with video). Gastrointest Endosc. 2023 Nov;98(5):755-764. doi: 10.1016/j.gie.2023.06.013. Epub 2023 Jun 24. PMID 37356632
- [Background] Masuelli L, Tumino G, Turriziani M, Modesti A, Bei R. Topical use of sucralfate in epithelial wound healing: clinical evidences and molecular mechanisms of action. Recent Pat Inflamm Allergy Drug Discov. 2010 Jan;4(1):25-36. doi: 10.2174/187221310789895649. PMID 19832693
- [Background] Ala S, Saeedi M, Janbabai G, Ganji R, Azhdari E, Shiva A. Efficacy of Sucralfate Mouth Wash in Prevention of 5-fluorouracil Induced Oral Mucositis: A Prospective, Randomized, Double-Blind, Controlled Trial. Nutr Cancer. 2016;68(3):456-63. doi: 10.1080/01635581.2016.1153666. Epub 2016 Mar 23. PMID 27007594